CLINICAL TRIAL: NCT03008811
Title: Norwegian Randomized Study of Persistent Atrial Fibrillation Treatment: Cryoballoon Versus Radiofrequency Catheter Ablation (NO PERS-AF)
Brief Title: Norwegian Study of Persistent Atrial Fibrillation Treatment: Cryoballoon Versus Radiofrequency Catheter Ablation
Acronym: NO PERS-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: St. Olavs Hospital (Other); University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/27
Record Dates: First submitted 2016-11-23; First posted 2017-01-02 (Estimated); Last update posted 2021-11-12 (Actual); Status verified 2020-02

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Atrial Fibrillation; Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cryoballoon (Active Comparator): Pulmonary vein isolation with cryoballoon catheter.
  Interventions: Procedure: Pulmonary vein isolation with cryoballoon catheter.
- Radiofrequency (Active Comparator): Pulmonary vein isolation with radiofrequency ablation catheter.
  Interventions: Procedure: Pulmonary vein isolation with radiofrequency ablation.

INTERVENTIONS:
Procedure: Pulmonary vein isolation with cryoballoon catheter. — Device: Arctic Front Advance™ cardiac cryoablation catheter system.
  Arms: Cryoballoon
Procedure: Pulmonary vein isolation with radiofrequency ablation. — Device: TactiCath™ Quartz irrigated ablation catheter (St. Jude Medical) with aid of 3-D mapping system (EnSite Precision, St. Jude Medical).
  Arms: Radiofrequency

SUMMARY:
This study will compare efficacy and safety of pulmonary vein isolation using a cryoballoon catheter versus a radiofrequency ablation with a contact force sensing catheter for treatment of patients with persistent or longstanding persistent atrial fibrillation.

DETAILED DESCRIPTION:
The purpose of this randomized clinical trial is to compare the efficacy and safety of pulmonary vein isolation with either the second generation cryoballoon (Arctic Front Advance™) or a radiofrequency ablation technique with an irrigated ablation catheter (TactiCath™ Quartz) . A total of 128 patients with persistent or longstanding persistent atrial fibrillation will be randomized for either radiofrequency or cryoballoon ablation treatment. With both techniques, pulmonary vein isolation will be performed and confirmed by a circular mapping catheter. The primary endpoint is freedom of any atrial arrhythmia recurrence at 12 months.Treatment success will be evaluated by using 12-lead electrocardiography and 7-day Holter recording.

ELIGIBILITY:
Inclusion criteria:

* Patients plan to undergo pulmonary vein isolation as the first procedure for symptomatic persistent atrial fibrillation (>7 days) and longstanding persistent atrial fibrillation (> 12 months, but ≤ 3 years) who are refractory to at least one class I or class III antiarrhythmic drug and required at least one electrical or pharmacologic cardioversion.
* Subject is at least 18 and ≤ 75 years old.
* Subject is able and willing to give informed consent.

Exclusion criteria:

* Subject has paroxysmal atrial fibrillation (< 7days) or persistent atrial fibrillation with duration > 3 years.
* Subject has any previous left atrial ablation procedure or surgery, including pulmonary vein isolation.
* Subject has presence of an intracavitary thrombus.
* Subject has uncontrolled heart failure.
* Subject has severe valvular disease.
* Subject has the left atrial diameter > 60 mm confirmed by echocardiography.
* Subject has contraindications to systemic anticoagulation with heparin or oral anticoagulants.
* Subject has known cryoglobulinaemia.
* Subject has severe renal dysfunction.
* Subject who is or may potentially be pregnant.
* Subject has unstable angina pectoris.
* Subject has history of previous myocardial infarction or percutaneous intervention during the last three months.
* Subject has chronic obstructive pulmonary disease with detected pulmonary hypertension.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
The freedom of any atrial arrhythmias at 12 months. | 12 months
  The primary endpoint is freedom of any atrial arrhythmias at 12 months (at least one episode of atrial fibrillation, or atrial flutter or atrial tachycardia with a duration > 30 seconds documented by 7-day Holter ECG, or any other printed ECG recording).

SECONDARY OUTCOMES:
Procedure duration | 12 months
  Procedure duration documented
Fluoroscopy time | 12 months
  Fluoroscopy time documented
Ablation time | 12 months
  Ablation time documented
Quality of life - Short Form (SF-36) Heath Survey | 12 months.
  Short Form (SF-36) Heath Survey filled in by patients.
Quality of life affected by atrial fibrillation. | 12 months.
  The Atrial Fibrillation Effect on Quality-of-life (AFEQT) questionnaire will be filled in by patients.
Admittance to hospital or emergency services due to symptoms caused by documented atrial arrhythmias. | 12 months.
  Hospitalization after the procedre
The burden of atrial fibrillation | 12 months.
  Total duration of atrial fibrillation recorded by 7-day Holter.
The occurrence of documented left atrial tachycardia and typical or atypical atrial flutter. | 12 months.
  Atrial tachycardia or atrial flutter recorded by all types of ECG
Symptoms related to atrial fibrillation. | 12 months.
  Symptoms related to atrial fibrillation documented
Serious adverse events. | 12 months.
  Serious adverse events documented

CONTACTS AND LOCATIONS:
Locations (3):
- Norway (3):
  - Haukeland University Hospital, Bergen
  - University Hospital of North Norway, Tromsø
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Camm AJ, Obel OA. Epidemiology and mechanism of atrial fibrillation and atrial flutter. Am J Cardiol. 1996 Oct 17;78(8A):3-11. doi: 10.1016/s0002-9149(96)00559-0. No abstract available. PMID 8903269
- [Background] Biblo LA, Yuan Z, Quan KJ, Mackall JA, Rimm AA. Risk of stroke in patients with atrial flutter. Am J Cardiol. 2001 Feb 1;87(3):346-9, A9. doi: 10.1016/s0002-9149(00)01374-6. PMID 11165976
- [Background] Vidaillet H, Granada JF, Chyou Po, Maassen K, Ortiz M, Pulido JN, Sharma P, Smith PN, Hayes J. A population-based study of mortality among patients with atrial fibrillation or flutter. Am J Med. 2002 Oct 1;113(5):365-70. doi: 10.1016/s0002-9343(02)01253-6. PMID 12401530
- [Background] Benjamin EJ, Wolf PA, D'Agostino RB, Silbershatz H, Kannel WB, Levy D. Impact of atrial fibrillation on the risk of death: the Framingham Heart Study. Circulation. 1998 Sep 8;98(10):946-52. doi: 10.1161/01.cir.98.10.946. PMID 9737513
- [Background] Wolf PA, Mitchell JB, Baker CS, Kannel WB, D'Agostino RB. Impact of atrial fibrillation on mortality, stroke, and medical costs. Arch Intern Med. 1998 Feb 9;158(3):229-34. doi: 10.1001/archinte.158.3.229. PMID 9472202
- [Background] Corley SD, Epstein AE, DiMarco JP, Domanski MJ, Geller N, Greene HL, Josephson RA, Kellen JC, Klein RC, Krahn AD, Mickel M, Mitchell LB, Nelson JD, Rosenberg Y, Schron E, Shemanski L, Waldo AL, Wyse DG; AFFIRM Investigators. Relationships between sinus rhythm, treatment, and survival in the Atrial Fibrillation Follow-Up Investigation of Rhythm Management (AFFIRM) Study. Circulation. 2004 Mar 30;109(12):1509-13. doi: 10.1161/01.CIR.0000121736.16643.11. Epub 2004 Mar 8. PMID 15007003
- [Background] Haissaguerre M, Jais P, Shah DC, Takahashi A, Hocini M, Quiniou G, Garrigue S, Le Mouroux A, Le Metayer P, Clementy J. Spontaneous initiation of atrial fibrillation by ectopic beats originating in the pulmonary veins. N Engl J Med. 1998 Sep 3;339(10):659-66. doi: 10.1056/NEJM199809033391003. PMID 9725923
- [Background] Verma A, Marrouche NF, Natale A. Pulmonary vein antrum isolation: intracardiac echocardiography-guided technique. J Cardiovasc Electrophysiol. 2004 Nov;15(11):1335-40. doi: 10.1046/j.1540-8167.2004.04428.x. PMID 15574190
- [Background] Oral H, Scharf C, Chugh A, Hall B, Cheung P, Good E, Veerareddy S, Pelosi F Jr, Morady F. Catheter ablation for paroxysmal atrial fibrillation: segmental pulmonary vein ostial ablation versus left atrial ablation. Circulation. 2003 Nov 11;108(19):2355-60. doi: 10.1161/01.CIR.0000095796.45180.88. Epub 2003 Oct 13. PMID 14557355
- [Background] Saad EB, Rossillo A, Saad CP, Martin DO, Bhargava M, Erciyes D, Bash D, Williams-Andrews M, Beheiry S, Marrouche NF, Adams J, Pisano E, Fanelli R, Potenza D, Raviele A, Bonso A, Themistoclakis S, Brachmann J, Saliba WI, Schweikert RA, Natale A. Pulmonary vein stenosis after radiofrequency ablation of atrial fibrillation: functional characterization, evolution, and influence of the ablation strategy. Circulation. 2003 Dec 23;108(25):3102-7. doi: 10.1161/01.CIR.0000104569.96907.7F. Epub 2003 Nov 17. PMID 14623799
- [Background] Pappone C, Rosanio S, Augello G, Gallus G, Vicedomini G, Mazzone P, Gulletta S, Gugliotta F, Pappone A, Santinelli V, Tortoriello V, Sala S, Zangrillo A, Crescenzi G, Benussi S, Alfieri O. Mortality, morbidity, and quality of life after circumferential pulmonary vein ablation for atrial fibrillation: outcomes from a controlled nonrandomized long-term study. J Am Coll Cardiol. 2003 Jul 16;42(2):185-97. doi: 10.1016/s0735-1097(03)00577-1. PMID 12875749
- [Background] Marrouche NF, Martin DO, Wazni O, Gillinov AM, Klein A, Bhargava M, Saad E, Bash D, Yamada H, Jaber W, Schweikert R, Tchou P, Abdul-Karim A, Saliba W, Natale A. Phased-array intracardiac echocardiography monitoring during pulmonary vein isolation in patients with atrial fibrillation: impact on outcome and complications. Circulation. 2003 Jun 3;107(21):2710-6. doi: 10.1161/01.CIR.0000070541.83326.15. Epub 2003 May 19. PMID 12756153
- [Background] Haissaguerre M, Jais P, Shah DC, Arentz T, Kalusche D, Takahashi A, Garrigue S, Hocini M, Peng JT, Clementy J. Catheter ablation of chronic atrial fibrillation targeting the reinitiating triggers. J Cardiovasc Electrophysiol. 2000 Jan;11(1):2-10. doi: 10.1111/j.1540-8167.2000.tb00727.x. PMID 10695453
- [Background] Ullah W, Hunter RJ, Haldar S, McLean A, Dhinoja M, Sporton S, Earley MJ, Lorgat F, Wong T, Schilling RJ. Comparison of robotic and manual persistent AF ablation using catheter contact force sensing: an international multicenter registry study. Pacing Clin Electrophysiol. 2014 Nov;37(11):1427-35. doi: 10.1111/pace.12501. Epub 2014 Sep 15. PMID 25220575
- [Background] Verma A, Jiang CY, Betts TR, Chen J, Deisenhofer I, Mantovan R, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P; STAR AF II Investigators. Approaches to catheter ablation for persistent atrial fibrillation. N Engl J Med. 2015 May 7;372(19):1812-22. doi: 10.1056/NEJMoa1408288. PMID 25946280
- [Background] Liu J, Kaufmann J, Kriatselis C, Fleck E, Gerds-Li JH. Second generation of cryoballoons can improve efficiency of cryoablation for atrial fibrillation. Pacing Clin Electrophysiol. 2015 Jan;38(1):129-35. doi: 10.1111/pace.12538. Epub 2014 Dec 12. PMID 25494851
- [Background] Jourda F, Providencia R, Marijon E, Bouzeman A, Hireche H, Khoueiry Z, Cardin C, Combes N, Combes S, Boveda S, Albenque JP. Contact-force guided radiofrequency vs. second-generation balloon cryotherapy for pulmonary vein isolation in patients with paroxysmal atrial fibrillation-a prospective evaluation. Europace. 2015 Feb;17(2):225-31. doi: 10.1093/europace/euu215. Epub 2014 Sep 3. PMID 25186456
- [Background] Ciconte G, Ottaviano L, de Asmundis C, Baltogiannis G, Conte G, Sieira J, Di Giovanni G, Saitoh Y, Irfan G, Mugnai G, Storti C, Montenero AS, Chierchia GB, Brugada P. Pulmonary vein isolation as index procedure for persistent atrial fibrillation: One-year clinical outcome after ablation using the second-generation cryoballoon. Heart Rhythm. 2015 Jan;12(1):60-6. doi: 10.1016/j.hrthm.2014.09.063. Epub 2014 Oct 2. PMID 25281891